CLINICAL TRIAL: NCT01833130
Title: Use of a Treatment Benefit Questionnaire in Patients With Chronic Migraine Treated With OnabotulinumtoxinA (BOTOX®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GMA-BTX-CM-12-545
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OnabotulinumtoxinA (Experimental): OnabotulinumtoxinA (botulinum toxin Type A) 155 units (U) total dose per treatment injected into specified head and neck muscles on Day 1 followed by a second treatment at Week 12.
  Interventions: Biological: OnabotulinumtoxinA
- Placebo (Normal saline) (Placebo Comparator): Placebo (Normal saline) injected into specified head and neck muscles on Day 1 followed by a second treatment at Week 12.
  Interventions: Drug: Normal saline (placebo)

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA (botulinum toxin Type A) 155 U total dose per treatment injected into specified head and neck muscles on Day 1 followed by a second treatment at Week 12.
  Other Names: botulinum toxin Type A; BOTOX®
  Arms: OnabotulinumtoxinA
Drug: Normal saline (placebo) — Placebo (Normal saline) injected into specified head and neck muscles on Day 1 followed by a second treatment at Week 12.
  Arms: Placebo (Normal saline)

SUMMARY:
This study will evaluate the use of the Assessment of Chronic Migraine Impacts (ACM-I) Questionnaire in assessing the impact and benefit of treatment with onabotulinumtoxinA (BOTOX®) in adults with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic migraine for at least 6 months prior to the screening visit
* Fifteen or more headache days during the 4-week screening period (≥4 headache episodes lasting ≥4 hours and ≥50 % of headache days are migraine)

Exclusion Criteria:

* Conditions causing chronic facial pain such as Temporomandibular Disorder (TMD) and fibromyalgia
* Use of headache prophylaxis medication within 4 weeks of the screening visit
* Diagnosis of Myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis
* Previous use of any botulinum toxin of any serotype for any reason
* Skin infections or acne that would interfere with the injection sites
* Acupuncture, transcutaneous electrical nerve stimulation (TENS), cranial traction, dental splints for headache, nociceptive trigeminal inhibition, occipital nerve block treatments, or injection of anesthetics/steroids within 4 weeks of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Safety Population includes all 52 patients who received at least one injection with the study treatment. The Intent-to-Treat (ITT) population consists of all 45 randomized patients. Seven (7) patients were excluded from the ITT population as they were withdrawn from the study due to a randomization error.
Period: Overall Study
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Started | 25 | 27
Completed | 15 | 8
Not Completed | 10 | 19

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population: all randomized patients (7 patients were withdrawn from the study due to a randomization error and excluded from the Intent-to-Treat population)
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 19 | 26 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (13.1) | 42.2 (11.8) | 42.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Assessment of Chronic Migraine Impacts (ACM-I) Questionnaire Total Score
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The total score ranged from 0 (lower impact chronic migraine) to 100 (highest impact chronic migraine). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 50.5 (17.6) | 47.2 (22)
  Change from Baseline at Week 24 (N=15, 18) | -25.2 (23.5) | -20.5 (24.6)

2. Secondary Outcome: Change From Baseline in the Symptom Severity Score (SSS) Subdomain of the Assessment of Chronic Migraine Symptoms (ACM-S) Questionnaire
Description: The ACM-S is 12 question migraine symptom scale over the past 24 hours. The SSS subdomain score ranges from 0 (no symptoms) to 100 (more severe symptoms). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the ACM-S SSS.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 54.3 (22.1) | 45.9 (25.9)
  Change from Baseline at Week 24 (N=14, 18) | -18.5 (39.2) | -17.5 (30.1)

3. Secondary Outcome: Change From Baseline in the Symptom Experience Score (SES) Subdomain of the ACM-S Questionnaire
Description: The ACM-S is 12 question migraine symptom scale over the past 24 hours. The SES subdomain score ranges from 0 (no symptoms) to 12 (all symptoms experienced). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the ACM-S SES.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 8.4 (2.6) | 8.2 (3.3)
  Change from Baseline at Week 24 (N=14, 18) | -1.6 (5.4) | -1.9 (5.1)

4. Secondary Outcome: Change From Baseline in the Activities of Daily Living Impact (ADL-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The ADL-I is a subdomain on the ACM-I. The ADL-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the ADL-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 45 (16.6) | 43.3 (21.1)
  Change from Baseline at Week 12 (N=15, 19) | -15.7 (24.7) | -15.3 (21.4)
  Change from Baseline at Week 22 (N=13, 15) | -30.4 (19.1) | -18.7 (24.4)
  Change from Baseline at Week 24 (N=15, 18) | -24 (24.8) | -21.9 (24.8)

5. Secondary Outcome: Change From Baseline in the Emotions Impact (EMO-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The EMO-I is a subdomain on the ACM-I. The EMO-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the EMO-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 51.9 (23.1) | 42.3 (25.4)
  Change from Baseline at Week 12 (N=15, 19) | -20 (32) | -13.9 (20.8)
  Change from Baseline at Week 22 (N=13, 15) | -26.7 (33.3) | -14.9 (26.6)
  Change from Baseline at Week 24 (N=15, 18) | -26.2 (28.4) | -16.3 (21)

6. Secondary Outcome: Change From Baseline in the Work/School Impact (WS-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The WS-I is a subdomain on the ACM-I. The WS-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the WS-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 47.9 (23.2) | 43.1 (26.9)
  Change from Baseline at Week 12 (N=15, 19) | -16.7 (36.4) | -20.5 (29.1)
  Change from Baseline at Week 22 (N=13, 15) | -32.3 (28.0) | -16 (40.7)
  Change from Baseline at Week 24 (N=15, 18) | -30 (28.0) | -18.9 (33.1)

7. Secondary Outcome: Change From Baseline in the Social Impact (SOC-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The SOC-I is a subdomain on the ACM-I. The SOC-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the SOC-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 39.6 (22.8) | 43.1 (26.3)
  Change from Baseline at Week 12 (N=15, 19) | -9.8 (25.7) | -21.8 (24.8)
  Change from Baseline at Week 22 (N=13, 15) | -19 (26.5) | -20 (28.4)
  Change from Baseline at Week 24 (N=15, 18) | -18.7 (25.5) | -19.6 (29.3)

8. Secondary Outcome: Change From Baseline in the Leisure Activities Impact (LEA-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The LEA-I is a subdomain on the ACM-I. The LEA-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the LEA-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 51.6 (21.4) | 55.4 (31.1)
  Change from Baseline at Week 12 (N=15, 19) | -16 (33.1) | -25.3 (27.4)
  Change from Baseline at Week 22 (N=13, 15) | -29.2 (24) | -22.7 (38.4)
  Change from Baseline at Week 24 (N=15, 18) | -26.7 (24.7) | -30.0 (37.7)

9. Secondary Outcome: Change From Baseline in the Household Activities Impact (HOS-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The HOS-I is a subdomain on the ACM-I. The HOS-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the HOS-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 45.3 (19.8) | 48.5 (23.4)
  Change from Baseline at Week 12 (N=15, 19) | -17.3 (30.1) | -18.9 (26.2)
  Change from Baseline at Week 22 (N=13, 15) | -27.7 (25.2) | -24 (34)
  Change from Baseline at Week 24 (N=15, 18) | -24 (28.5) | -24.4 (29.6)

10. Secondary Outcome: Change From Baseline in the Energy Impact (ENE-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The ENE-I is a subdomain on the ACM-I. The ENE-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the ENE-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 58.2 (22.2) | 60.2 (19.9)
  Change from Baseline at Week 12 (N=15, 19) | -19.7 (34.2) | -22.4 (24.1)
  Change from Baseline at Week 22 (N=13, 15) | -33.1 (30.3) | -20 (31.8)
  Change from Baseline at Week 24 (N=15, 18) | -26.3 (27.3) | -23.3 (27.8)

11. Secondary Outcome: Change From Baseline in the Cognitive Impact (COG-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The COG-I is a subdomain on the ACM-I. The COG-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the COG-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 18 | 26
Scores on a Scale
  Baseline | 60.0 (19.9) | 52.6 (27.0)
  Change from Baseline at Week 12 (N=15, 19) | -25.2 (29.8) | -20.7 (25.5)
  Change from Baseline at Week 22 (N=13, 15) | -31.1 (30.3) | -20.9 (32.8)
  Change from Baseline at Week 24 (N=14, 18) | -31.8 (29.3) | -26.3 (27.3)

12. Secondary Outcome: Change From Baseline in the General Impact (GEN-I) Domain of the ACM-I Questionnaire
Description: The ACM-I is a 24 question scale used to measure the impact of chronic migraine on daily activities and patient-treatment benefit over the past 7 days. The GEN-I is a subdomain on the ACM-I. The GEN-I score ranged from 0 (lowest impact) to 100 (highest impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the GEN-I.
Time Frame: Baseline, Week 12, Week 22, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 57.9 (23) | 53.1 (29.9)
  Change from Baseline at Week 12 (N=15, 19) | -22.7 (36.1) | -18.9 (25.4)
  Change from Baseline at Week 22 (N=12, 15) | -38.3 (31.3) | -10.7 (39.2)
  Change from Baseline at Week 24 (N=14, 18) | -28.6 (31.1) | -15.6 (45.3)

13. Secondary Outcome: Change From Baseline in the Headache Impact Test-6 (HIT-6) Questionnaire Total Score
Description: The HIT-6 is a 6 question 5-point scale used to measure the impact of headaches on daily life. The total score ranged from 36 (no impact) to 78 (worst impact). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 64.7 (4.2) | 65.3 (5.5)
  Change from Baseline at Week 24 (N=15, 18) | -5.1 (4.7) | -6.7 (7.9)

14. Secondary Outcome: Change From Baseline in the Role Function-Restrictive (RR) Domain of the Migraine Specific Questionnaire (MSQ)
Description: The MSQ is 14 question scale that measures health-related impairments attributed to migraines over the past 4 weeks. The RR domain score ranges from 0 (no symptoms) to 100 (symptoms experienced all the time). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the RR.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 39.8 (16.6) | 40.9 (21.7)
  Change from Baseline at Week 24 (N=13, 18) | 32.1 (15.4) | 26.5 (28.9)

15. Secondary Outcome: Change From Baseline in the Role Function-Preventive (RP) Domain of the MSQ
Description: The MSQ is 14 question scale that measures health-related impairments attributed to migraines over the past 4 weeks. The RP domain score ranges from 0 (no symptoms) to 100 (symptoms experienced all the time). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the RP.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 58.9 (18.8) | 62.5 (23.0)
  Change from Baseline at Week 24 (N=13, 18) | 25.8 (18) | 20.8 (28.9)

16. Secondary Outcome: Change From Baseline in the Emotional Function (EF) Domain of the MSQ
Description: The MSQ is 14 question scale that measures health-related impairments attributed to migraines over the past 4 weeks. The EF domain score ranges from 0 (no symptoms) to 100 (symptoms experienced all the time). A negative number change from baseline indicates an improvement, and a positive number change from baseline indicates a worsening in the EF.
Time Frame: Baseline, Week 24
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 26
Scores on a Scale
  Baseline | 53.3 (27.6) | 58.7 (23.9)
  Change from Baseline at Week 24 (N=14, 18) | 26.2 (26.3) | 18.5 (34.2)

ADVERSE EVENTS:
Description: The Safety Population is used to assess adverse events (AEs) and serious adverse events (SAEs) and includes all subjects who received at least one study treatment injection.
Arm/Group | OnabotulinumtoxinA | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/27
Other Adverse Events (participants affected / at risk) | 9/25 | 2/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA (N=25) | Placebo (Normal Saline) (N=27)
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA (N=25) | Placebo (Normal Saline) (N=27)
Injection Site Pain (General disorders) | 2 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Facial Paresis (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.